CLINICAL TRIAL: NCT02984085
Title: Prospective, Open-label, Uncontrolled Clinical Trial to Assess the Safety and Efficacy of Autologous Cultured Epidermal Grafts Containing Epidermal Stem Cells Genetically Modified With a Gamma-retroviral (rv) Vector Carrying COL7A1 cDNA for Restoration of Epidermis in Patients With Recessive Dystrophic Epidermolysis Bullosa.
Brief Title: Clinical Trial to Assess Safety and Efficacy of Autologous Cultured Epidermal Grafts Containing Epidermal Stem Cells Genetically Modified in Patients With RDEB.
Acronym: HOLOGENE7
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Replaced by new study in progress
Sponsor: Holostem s.r.l. (Industry)
Collaborators: Paracelsus Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOLOGENE 7
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Recessive Dystrophic Epidermolysis Bullosa
Keywords: RDEB; Stem cells; Gene therapy
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica | interventions — cyclic adenosine-5'-trimetaphosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Genetically corrected cultured epidermal autograft (Experimental): The surgery will be carried out in 2 stages, the first aims at taking biopsy to isolate epidermal cells including stem cells. The biopsy will be processed in a laboratory of a regenerative medicine manufacturing site where they will be corrected, expanded and prepared as final sheets to be implanted.
  In the second surgery, genetically corrected cultured epidermal autograft (Hologene 7) will be implanted into the selected area. The specialist surgeon will either use a local or general anaesthetic for the implant operation. The treated area will be immobilized for some days after this operation. Antibiotics and anti-inflammatory drugs will be administered (if necessary) to prevent infections and to minimise swelling.
  Interventions: Drug: Genetically corrected cultured epidermal autograft (ATMP)

INTERVENTIONS:
Drug: Genetically corrected cultured epidermal autograft (ATMP) — Genetically corrected cultured epidermal autograft (Hologene 7) is intended for transplantation onto surgically prepared blistering skin areas of RDEB patients and permanent regeneration of a healthy, functional and renewing epidermis sustained by the engraftment of transduced epidermal stem cells.
  By taking some autologous epidermal cells, a new layer of transgenic tissue is grown in the laboratory. This layer of tissue is then implanted by a surgeon into the damaged area. The implantation can be done in one or more areas and repeated in case of failure of the first surgery.
  Other Names: Hologene 7 Study product (ATMP)

SUMMARY:
Prospective open-label, uncontrolled clinical study to assess the safety and efficacy of autologous cultured epidermal grafts containing epidermal stem cells genetically modified with the aid of a gamma-retroviral vector carrying COL7A1 complementary DNA (cDNA) for restoration of the epidermis in patients with recessive dystrophic epidermolysis bullosa. The purpose of this study is to demonstrate the safety and efficacy after one or more treatments with genetically corrected cultured epidermal autograft (Hologene 7) in patients suffering of recessive dystrophic epidermolysis bullosa (RDEB) with COL7A1 mutation.

DETAILED DESCRIPTION:
This is a monocentric, prospective, open label, uncontrolled clinical trial, phase I/II.

Patients will be screened according to the Study Inclusion and Exclusion criteria and will be candidate for the treatment if all inclusion and none of the exclusion criteria are met.

After confirmation of eligibility, patients will undergo biopsy for the collection of the autologous epidermal cells to be used to produce the tissue for the treatment. In case all criteria are met, the transplantation of the new cultured transgenic epidermis will be planned according to the procedures and the need of the patient.

The study treatment consists of a surgical intervention for new restored stem cells implantation.

The surgery will be carried out in 2 stages, the first aims at taking biopsy to isolate epidermal cells including stem cells. The biopsy will be processed in a laboratory of a regenerative medicine manufacturing site where they will be corrected, expanded and prepared as final sheets to be implanted. Therefore, the patient can have his second intervention. In this second surgery, genetically corrected cultured epidermal autograft (Hologene 7) will be implanted into the selected area. The specialist surgeon will either use a local or general anaesthetic for the implant operation. The treated area will be immobilized for some days after this operation. Antibiotics and anti-inflammatory drugs will be administered (if necessary) to prevent infections and to minimise swelling.

Three months after the transplantation, primary endpoint will be evaluated by the Investigator. The study completion will be reached when 1 year (secondary endpoint) of follow-up after the last transplant in the last patient will be accomplished.

The end of the trial is defined as the last visit of the last patient after the last treatment if any.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent prior to any study-related procedures. Informed consent will also include the possibility of additional transplantations and of the rolling over to the long-term extension period;
2. Adult male and female patients (≥18 years old and < 55); Paediatric patients aged 6 to 17 years will be also enrolled.
3. RDEB molecular characterization by mutation analysis;
4. Non-collagenous domain (NC1 or NC2) antibody immunofluorescence or staining positive in Western Blot;
5. Presence of chronic (persistent for more than 3 months) large wounds (>10 cm2) and/or erosion;
6. A cooperative attitude to follow up the study procedures (Caregivers in case of minors).

Exclusion Criteria:

1. Known or suspected intolerances against anaesthesia;
2. Bad general condition (ECOG index >1)
3. Unresectable or metastasizing squamous cell carcinoma (SCCs);
4. Antibodies to type VII collagen associated antigens demonstrated on indirect immunofluorescence;
5. Clinical and/or laboratory signs of acute systemic infections at the time of screening. Patient can be re-screened after appropriate treatment;
6. Severe systemic diseases (i.e. uncompensated diabetes);
7. Female subjects: pregnant or lactating women and all women physiologically capable of becoming pregnant (i.e. women of childbearing potential) UNLESS they are willing to use one or more reliable methods of contraception with a Pearl index ≤1.
8. Allergy, sensitivity or intolerance to drugs or excipients (hypersensitivity to any of the excipients listed in Investigator's brochure or in this protocol):

   * Transport medium (Dulbecco's Modified Eagles Medium supplemented with L-glutamine)
   * Fibrin support
   * Betaisodona
9. Contraindications to the local or systemic antibiotics and/ or corticosteroids foreseen by the protocol;
10. Contraindications to undergo extensive surgical procedures;
11. Clinically significant or unstable concurrent disease or other clinical contraindications to stem cell transplantation based upon investigator's judgment or other concomitant medical conditions affecting grafting procedure;
12. Patients (or parents in case of paediatric subject) unlikely to comply with the study protocol or unable to understand the nature and scope of the study or the possible benefits or unwanted effects of the study procedures and treatments.
13. Participation in another clinical trial where investigational drug was received less than 6 months prior to screening visit.

Ages: 6 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2018-08-06 (Actual); Study Completion 2018-08-06 (Actual)

PRIMARY OUTCOMES:
Safety | 3-month
  number and percentage of patients experiencing treatment-related adverse events (TRAEs), serious adverse events (SAEs) and serious adverse drug reactions (ADRs) up to 3 months after the first treatment.

SECONDARY OUTCOMES:
Efficacy | 3- and 12-months
  Percentage of patients with clinical success after one or more treatments with study product at 3 and 12 months follow up.
  Clinically success is reached when both the following conditions are met:
  o Regeneration of a clinically normal appearing skin with absence of detectable blister.
  AND
  o Restoration of type VII collagen expression and restoration of anchoring fibrils in the treated area.

OTHER OUTCOMES:
Treatment success | 12-months
  Percentage of patients defined as "success" by Investigator site according to the same parameters as for the primary and key secondary efficacy assessments 12 months after last treatment;
Fibrin re-absorption | 1- and 4-weeks
  • Complete matrix re-absorption (by visual inspection) one week after the transplantation and clinical success (defined as the primary efficacy assessment) at early assessment time points (1 and 4 weeks after transplantation).

CONTACTS AND LOCATIONS:
Overall Officials: Michele De Luca, MD/Professor, Study Director — Holostem s.r.l.; Johann W. Bauer, MD, Principal Investigator — Paracelsus Medical University - EB House
Locations (1):
- EB House Austria, Department of Dermatology, Paracelsus Medical University, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Correction of junctional epidermolysis bullosa by transplantation of genetically modified epidermal stem cells. — https://www.ncbi.nlm.nih.gov/pubmed/17115047
- See also: Long-term stability and safety of transgenic cultured epidermal stem cells in gene therapy of junctional epidermolysis bullosa. — https://www.ncbi.nlm.nih.gov/pubmed/24511464
- See also: Closure of a large chronic wound through transplantation of gene-corrected epidermal stem cells. — https://www.ncbi.nlm.nih.gov/pubmed/27840234